CLINICAL TRIAL: NCT00003578
Title: A Randomized Trial to Evaluate Early High Dose Therapy and Autologous Bone Marrow Transplantation as Part of Planned Initial Therapy for Poor Risk Intermediate/High Grade NHL
Brief Title: High Dose Chemotherapy With or Without Bone Marrow Transplantation in Treating Patients With Intermediate- or High-Grade Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lymphoma Trials Office (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066645; BNLI-LY02; EU-98039
Record Dates: First submitted 1999-11-01; First posted 2004-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2007-05

CONDITIONS: Lymphoma
Keywords: stage III grade 3 follicular lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic | interventions — VAP-cyclo protocol; Carmustine; Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide; Melphalan; Prednisone; Vincristine; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: CHOP regimen
Drug: carmustine
Drug: cyclophosphamide
Drug: cytarabine
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: melphalan
Drug: prednisone
Drug: vincristine sulfate
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Bone marrow transplantation may allow doctors to give higher doses of chemotherapy drugs and kill more cancer cells. It is not yet known whether high dose chemotherapy plus bone marrow transplantation is more effective than high dose chemotherapy alone for intermediate- or high-grade non-Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of high dose chemotherapy with or without bone marrow transplantation in treating patients who have intermediate- or high-grade non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the value of early intensification with autologous bone marrow transplantation or stem cell support in patients with poor prognosis intermediate or high grade non-Hodgkin's lymphoma.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by age (under 50 vs 50 and over), bone marrow involvement (yes vs no), and country. All patients receive cyclophosphamide, doxorubicin, and vincristine on day 1 and prednisone on days 1-5. Courses repeat every 21 days. Patients receive a minimum of 6 courses of treatment in the absence of disease progression and unacceptable toxicity. Arm I: Patients receive carmustine IV over 2 hours on day 1 in week 9 or 10. Etoposide and cytarabine IV are administered over 30 minutes on days 2-5. Melphalan IV is administered over 5 minutes on day 6. Patients receive cryopreserved bone marrow or peripheral blood stem cells on day 7. Arm II: Patients continue conventional therapy. Patients are followed at 8-9 weeks and 6 months.

PROJECTED ACCRUAL: This study will accrue 500 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed intermediate or high grade adult non-Hodgkin's lymphoma: Follicular large cell lymphoma Diffuse mixed cell lymphoma Diffuse large cell lymphoma Diffuse immunoblastic lymphoma Poor prognostic features defined as the presence of 2 or 3 of the following: Stage III/IV Lactase dehydrogenase greater than normal ECOG performance status 2-4 A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 16 to 65 Performance status: See Disease Characteristics Life expectancy: Not specified Hematopoietic: Not specified Hepatic: See Disease Characteristics Renal: Not specified Other: No other medical condition prohibiting intensive therapy

PRIOR CONCURRENT THERAPY: At least 5 years since prior systemic therapy for cancer

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 1993-01

CONTACTS AND LOCATIONS:
Overall Officials: David C. Linch, Study Chair — University College London Hospitals
Locations (72):
- Charles University Hospital, Prague (Praha), Czechia
- Denmark (2):
  - Aarhus Amtssygehus, Aarhus
  - Rigshospitalet, Copenhagen
- Norway (3):
  - Norwegian Radium Hospital, Oslo
  - Ullevall Hospital, Oslo
  - University of Tromso, Tromsø
- United Kingdom (66):
  - Stoke Mandeville Hospital, Aylesbury-Buckinghamshire, England
  - Royal United Hospital, Bath, England
  - City Hospital - Birmingham, Birmingham, England
  - Birmingham Heartlands and Solihull NHS Trust (Teaching), Birmingham, England
  - Southmead Hospital, Bristol, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Queen's Hospital, Burton, Burton-on-Trent, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Cheltenham General Hospital, Cheltenham, England
  - Countess of Chester Hospital, Chester, England
  - Derbyshire Royal Infirmary, Derby, England
  - Royal Free Hospital, Hampstead, London, England
  - Northwick Park Hospital, Harrow, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Ipswich Hospital NHS Trust, Ipswich, England
  - Leeds Teaching Hospital Trust, Leeds, England
  - University Hospitals of Leicester, Leicester, England
  - Royal Liverpool and Broadgreen Hospitals, Liverpool, England
  - Whipps Cross Hospital, London, England
  - Saint Bartholomew's Hospital, London, England
  - St. Bartholomew's Hospital, London, England
  - St. Georges Hospital Medical School, London, England
  - University College London Medical School, London, England
  - University College London, London, England
  - Charing Cross Hospital, London, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Southport and Formby District General Hospital, Merseyside, England
  - Milton Keynes General Hospital, Milton Keynes, England
  - Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Derriford Hospital, Plymouth, England
  - Oldchurch Hospital, Romford, England
  - Pembury Hospital, Royal Tunbridge Wells, Kent, England
  - Sheffield Teaching Hospitals, Sheffield, England
  - Weston Park Hospital, Sheffield, England
  - Royal South Hants Hospital, Southampton, England
  - Royal Marsden Hospital, Sutton, England
  - Torbay Hospital, Torquay Devon, England
  - Hillingdon Hospital, Uxbridge, England
  - Sandwell District General Hospital, West Bromwich, England
  - Good Hope Hospital Trust, West Midlands, England
  - Pontefract General Infirmary, West Yorks, England
  - New Cross Hospital, Wolverhampton, England
  - Belfast City Hospital Trust, Belfast, Northern Ireland
  - Altnagelvin Area Hospital, Londonderry, Northern Ireland
  - Ysbyty Gwynedd, Bangor, Wales
  - Royal Bournemouth Hospital, Bournemouth
  - Law Hospital, Carluke UK
  - Saint Richards Hospital, Chichester
  - Chase Farm Hospital, Enfield
  - Epsom General Hospital, Epsom Surrey
  - Grantham and District Hospital, Grantham
  - King George Hospital, Ilford, Essex
  - Queen Elizabeth Hospital, Kings Lynn
  - Walton General Hospital, Liverpool
  - Newham General Hospital, London
  - St. Mary's Hospital, London
  - West Middlesex Hospital, Middlesex
  - East Surrey Hospital, Redhill
  - Rotherham District General Hospital-NHS Trust, Rotherham
  - Scunthorpe General Hospital, Scunthorpe
  - Staffordshire General Hospital, Stafford